CLINICAL TRIAL: NCT05873517
Title: Pragmatic, Waitlist Randomized Controlled Trial of a Trauma-Focused Intervention With Women Experiencing Homelessness
Brief Title: Trauma-Focused Intervention With Women Experiencing Homelessness
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Principal Investigator left the institution
Sponsor: Rush University Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22060903-IRB01
Record Dates: First submitted 2023-04-12; First posted 2023-05-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Psychological Trauma; Trauma and Stress Related Disorders; Substance-Related Disorders; Substance Use; Substance Use Disorders
Keywords: Homelessness
MeSH Terms: conditions — Psychological Trauma; Trauma and Stressor Related Disorders; Substance-Related Disorders | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Eligible participants will either receive immediate NET+ or be assigned to a waitlist; all participants will be offered the opportunity to enroll in the NET+ intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate NET+ (Experimental): Receives NET+ immediately
  Interventions: Behavioral: Immediate Narrative Exposure Therapy (NET)+
- Waitlist NET+ (Active Comparator): Receives NET+ after waitlist
  Interventions: Behavioral: Waitlist + NET+

INTERVENTIONS:
Behavioral: Immediate Narrative Exposure Therapy (NET)+ — The basis of this intervention is adapted Narrative Exposure Therapy (NET)+. All participants receive 4-8 active NET+ sessions, including a psychoeducational session.
  Arms: Immediate NET+
Behavioral: Waitlist + NET+ — Waitlist control group participants receive 1 psychoeducational sessions and will be added to a waitlist; waitlist control group participants randomly selected from the waitlist be offered the opportunity to receive the active intervention (NET+).
  Arms: Waitlist NET+

SUMMARY:
Homelessness and associated traumas disproportionately affect women. The biopsychosocial health consequences of untreated trauma are profound. PTSD frequently co-occurs with other chronic health conditions, including substance use disorders (SUD). Co-morbid PTSD and SUD (PTSD+SUD) is common and difficult to treat, resulting in severe morbidity and premature mortality among women experiencing homelessness. Executing this study will help to address the disproportionate PTSD+SUD comorbidity burden, which drives health inequities in the growing population of women experiencing homelessness within and beyond Chicago.

DETAILED DESCRIPTION:
Homelessness and associated traumas disproportionately affect women. The biopsychosocial health consequences of untreated trauma are profound. PTSD frequently co-occurs with other chronic health conditions, including substance use disorders (SUD). Co-morbid PTSD and SUD (PTSD+SUD) is common and difficult to treat, resulting in severe morbidity and premature mortality among women experiencing homelessness. We have systematically adapted a trauma-focused intervention protocol (Narrative Exposure Therapy [NET]) to the self-identified needs and preferences of trauma-affected women experiencing homelessness. This adapted intervention, "NET+", incorporates strengths and preferences identified by women themselves, embedding principles of cognitive behavioral therapy (CBT) into conventional NET. NET+ aims to both employ core NET principles to re-process past trauma in parallel with building present-centered skills to address avoidant coping motives in PTSD+SUD. Via a pragmatic, waitlist randomized controlled trial, we will further assess the feasibility, acceptability, and preliminary effects of a 3-week NET+ intervention protocol with up to 100 women experiencing homelessness. We will determine pre- and post-NET+ intervention PTSD and trauma-related symptom scores (depression, anxiety, somatization, sleep), substance use behaviors, and effect sizes. Executing this study will help to address the disproportionate PTSD+SUD comorbidity burden, which drives health inequities in the growing population of women experiencing homelessness within and beyond Chicago.

ELIGIBILITY:
Inclusion Criteria:

* self-identifies as a woman;
* greater than or equal to 18 years;
* positive screen on TAPS-1 (reflecting problematic substance use);
* recently (within 1 year) or currently homeless (HRSA definition);
* affected by a traumatic life event and trauma-related distress (+Life Events Checklist for DSM-5 Standard [LEC-5] response ≥1 and PTSD Checklist for DSM-5 [PCL-5] score ≥28).

Exclusion Criteria:

- impaired decisional capacity to consent to participation (University of California, San Diego Brief Assessment of Capacity to Consent [UBACC] score ≤14.5)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identifies as "woman"
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder Symptoms | 6 weeks
  PTSD Checklist for DSM-5 (PCL-5), range 0-80, higher scores = worse outcome

SECONDARY OUTCOMES:
Depression | 6 weeks
  Patient Health Questionnaire-9, range 0-27, higher scores = worse outcome
Anxiety | 6 weeks
  Generalized Anxiety Disorder 7-item (GAD-7), range 0-27, higher scores = worse outcome
Sleep Problems | 6 weeks
  Insomnia Severity Index (ISI), range 0-28, higher scores = worse outcome
Substance Use | 6 weeks
  Tobacco, Alcohol, Prescription substance use behaviors, medication, and other Substance use Tool (positive/negative screen - positive screen = using substances/worse outcomes)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Deborah's Place, Chicago, Illinois
  - Sarah's Circle, Chicago, Illinois